CLINICAL TRIAL: NCT02734498
Title: Prospective Treatment Study of Catatonia Patients With Right Unilateral Electroconvulsive Treatment (RUL ECT) and Bilateral Electroconvulsive Treatment (BL ECT) Regimens
Brief Title: Prospective Treatment Study of Catatonia Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00031669
Record Dates: First submitted 2016-03-23; First posted 2016-04-12 (Estimated); Results first posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Catatonia
MeSH Terms: conditions — Catatonia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Right unilateral (RUL) ECT (Active Comparator): Right Unilateral placement of treatment electrodes in electroconvulsive treatment.
  Interventions: Device: Electroconvulsive Treatment (ECT) Right Unilateral
- Bilateral (BL) ECT (Active Comparator): Bilateral placement of treatment electrodes in electroconvulsive treatment.
  Interventions: Device: Electroconvulsive Treatment (ECT) - Bilateral
- Control group (No Intervention): No ECT treatment for control group.

INTERVENTIONS:
Device: Electroconvulsive Treatment (ECT) Right Unilateral — Intervention is electroconvulsive treatment (ECT) involves a brief electrical stimulation of the brain while the patient is under anesthesia. Performed unilateral on the right side.
  Arms: Right unilateral (RUL) ECT
Device: Electroconvulsive Treatment (ECT) - Bilateral — Intervention is electroconvulsive treatment (ECT) involves a brief electrical stimulation of the brain while the patient is under anesthesia. Performed Bilateral.
  Arms: Bilateral (BL) ECT

SUMMARY:
The purpose of this treatment study is to compare the effectiveness of different electrode placements used in Electroconvulsive Therapy (ECT) in the treatment of catatonia. In this study Electroconvulsive Therapy will be compared to medications used in the treatment of catatonia. Medications will be administered by the primary team as part of standard of care. Medications are not primarily being used as a part of this research study.

This treatments study, will be able to compare response rate of catatonia to right unilateral electroconvulsive treatment (RUL ECT) and Bilateral electroconvulsive treatment (BL ECT). Also having a control group of catatonia patients, which will not be treated with ECT will provide additional information on early ECT treatment of Catatonia.

DETAILED DESCRIPTION:
Catatonia was first described in 1873 by a German psychiatrist, Karl Ludwig Kahlbaum in his monograph titled ''Die Katatonie oder Das Spannungsirresein'' (Catatonia or tension insanity) (Kahlbaum, 1873). He conceptualized catatonia as a motor syndrome characterized by lack of motion, speech, alternating with periods of excessive purposeful motor activity, rigidity, negativism, verbigeration, automatic imbalance, posturing, grimacing and stereotypes. He also described that the syndrome generally had a periodic course and lethal outcome in a few. Despite a long history, "katatonia" was associated with different illnesses and was given as diagnostic specifier. DSM- V made a change and added catatonia as an independent diagnostic symptom.

According to DSM-V, catatonia is characterized by the following:

A. the clinical picture is dominated by 3 or more of the following symptoms

(1) Stupor (2) Catalepsy (3) Waxy flexibility (4) Mutism (5) Negativism (6) Posturing (7) Mannerism (8) Stereotypy (9) Agitation (10) Grimacing (11) Echolalia (12) Echopraxia

B. There is evidence from the history, physical examination or laboratory findings that the disturbance is in the direct patho-physiological consequence of another medical condition.

C. The disturbance is not better explained by another mental disorder

D. the disturbance does not occur exclusively during the course of a delirium

E. The disturbance causes clinically significant distress or impairment in social, occupational or other important areas of functioning

Electroconvulsive therapy has a very good track record in treatment of catatonia (World J Psychiatr. 2015 June 22; 5(2): 182-192), but current literature does not shed light on the speed and degree of response of catatonia to ECT. This study aims to analyze and describe the change of clinical signs and symptoms as a response parameter to judge ECT treatment series efficacy.

This treatment study, will be able to compare response rate of catatonia to right unilateral electroconvulsive treatment (RUL ECT) and Bilateral electroconvulsive treatment (BL ECT). Also having a control group of catatonia patients, which will not be treated with ECT will provide additional information on early ECT treatment of Katatonia.

Objectives:

1. To study the response rate of catatonia to right unilateral (RUL) ECT and bilateral (BL) ECT.
2. To compare response rate of catatonia to RUL ECT and BL ECT
3. To analyze and describe the change of clinical signs and symptoms after ECT treatment series

Methods and Measures:

Design This study is a case control study. Currently ECT is considered standard of treatment for catatonia in addition to alternative medication options.

Study participants meeting inclusion and exclusion criteria will be and providing informed consent will be randomly assigned to receive either bilateral electroconvulsive treatment (BL ECT) or right unilateral electroconvulsive treatment (RUL ECT).

* Patients who are otherwise eligible and consent to participate in our study, but refuse ECT (or ones who are unable to consent but their court appointed legal guardian or health care power of attorney refuse ECT) will be enrolled as a control group. The control group will undergo all the same laboratory investigations and Bush Francis measurements for evaluation of their catatonia but will not receive ECT.
* Informed consent will be obtained from the study participant or their legally authorized representative by the principal investigator or sub-investigator.
* Prior to treatment each patient will be examined by a clinician (psychiatrist and psychiatric resident) in which the following information will be obtained:

  1. Psychiatric interview with uniformed questioner
  2. History of the present illness (HPI) with onset, course of presenting symptoms, comorbidities, precipitating illness or life events - emphasis upon psychological stress
  3. Substance abuse screening
  4. Psychiatric history - Psychiatric diagnoses with age/date of diagnoses
  5. Medical history, with focus on comorbid developments and chronic medical disease states - especially if recent worsening or change in therapy
  6. Previous episodes of catatonia - dates and pertinent developments to social history (as noted above with HPI) with time course and treatment response/failure to ECT or medications
  7. Recent medication changes, with specific focus on timing of symptoms if possible - regimen prior to symptom/sign development, medication changes, and current medication
  8. Neurological conditions - including Traumatic brain injury (TBI), seizure history, neurodevelopmental disorders, delirium, dementia. The Montreal Cognitive Assessment (MOCA) will be administered the day prior to each ECT treatment and the day after each ECT treatment for pre and post procedure cognitive monitoring.
  9. Incontinence
  10. Medical, metabolic, and/or psychiatric comorbidities are recorded but intentionally NOT excluded, with limited exceptions:Cerebrovascular accident (CVA).
  11. Questionnaires and rating scales: The following instruments will be administered by a trained clinician (psychiatric resident, medical student):

      1. Bush- Francis Scale (BFCRS): The BFCRS is a rating scale consisting of 23 catatonia items (Bush et al., 1996a). The first 14 items on this scale are the most common, classical sings of catatonia & are also known as Catatonia Screening Instrument (BFCSI). If two or more of the BFCSI signs are present, for 24 hours or longer, catatonia is a possibility (Sienaert et al, 2011). For the purpose of this study, a score of 4 or more on the 23-item BCFRS will be considered for inclusion in this study.
      2. Hamilton depression scale
      3. Montreal Cognitive Assessment (MoCA)

      The administration of the BFCRS, Hamilton depression scale and MoCA will be videotaped for additional rating by a blinded rater. These assessments will be administered before and after each ECT treatment.
  12. Labs and testing to rule out organic causes of catatonia include:

      EEG electroencephalogram EKG - electrocardiogram CT scan of the head w/o contrast CMP complete metabolic panel, CBC diff complete blood count with differential Thyroid studies TSH T3 T4 Metabolic/Inflammatory laboratory tests (in specific conditions) Urine Analysis with Urine Drug Screen within 48 hours of admission) Fe serum level Fibrin D-dimer Magnesium (Mg)
  13. Pre-anesthesia work-up performed by the department of anesthesia to determine fitness for ECT. Anesthesia faculty will administer anesthesia to participants during the ECT procedure. They will monitor patient in the operating room (OR) before, during and after the ECT procedure for at least 30 minutes for any adverse effects.
  14. ECT treatments will begin after initial evaluation as described above. ECT treatments will be administered three times a week.
  15. Participants will not be required to try and fail a challenge of Intravenous (IV) or Intramuscular (IM) Lorazepam prior to being assigned to receive ECT treatments.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to WFBMC Inpatient Psychiatry unit with catatonia who are clinically eligible for ECT.
* Clinical catatonia as evidenced by a Bush-Francis Catatonia Rating Scale (BFCRS) score of 4 or more

Exclusion Criteria:

* Pregnant women

Patients with any of the following medical conditions which are contraindications for ECT:

* Pheochromocytoma
* History of stroke within the past 3 months
* Cardiac conduction defects
* Cerebral or aortic aneurysms

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-01; Primary Completion 2017-03-19 (Actual); Study Completion 2017-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Kimball, M.D, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Personal data of psychiatric patients will not be shared.

RESULTS

PARTICIPANT FLOW:
Groups:
- Right Unilateral (RUL) ECT: Right Unilateral placement of treatment electrodes in electroconvulsive treatment.
  Electroconvulsive Treatment (ECT): Intervention is electroconvulsive treatment (ECT) involves a brief electrical stimulation of the brain while the patient is under anesthesia
- Bilateral (BL) ECT: Bilateral placement of treatment electrodes in electroconvulsive treatment.
  Electroconvulsive Treatment (ECT): Intervention is electroconvulsive treatment (ECT) involves a brief electrical stimulation of the brain while the patient is under anesthesia
Period: Overall Study
Arm/Group | Right Unilateral (RUL) ECT | Bilateral (BL) ECT | Control Group
Started | 2 | 0 | 0
Completed | 2 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study design was too complicated and therefore too difficult to enroll. The study team was unable to continue recruiting because of lack of resources.
Groups:
- Total: Total of all reporting groups
Arm/Group | Right Unilateral (RUL) ECT | Bilateral (BL) ECT | Control Group | Total
Number analyzed (Participants) | 2 | 0 | 0 | 2
Age, Customized [Number; unit: participants] — Age not collected to protect patient confidentiality since there are only two
  participants
    not collected | 2 |  |  | 2
Sex/Gender, Customized [Count of Participants; unit: Participants] — not collected to protect PHI since there were only two participants
  Participants
    Not collected | 2 |  |  | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 2 |  |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Catatonia on the Bush- Francis Scale (BFCRS) - Pre
Description: Repetitive evaluation by the Bush- Francis Scale (BFCRS) - To assess excitement, immobility, mutism, staring, posturing/catalepsy, grimacing, echopraxia, stereotypy, mannerisms, verbigeration, rigidity, negativism, waxy flexibility, withdrawal, impulsivity, automatic obedience, mitgehen, gegenhalten, ambitendency, grasp reflex, preservation, combativeness and automatic abnormality. Contains 23 items rated using a scale of 0-3. Total Score 0-69. Higher scores denote worse outcomes.
Time Frame: Prior first ECT treatment
Population: Only two participants enrolled because study ended. Both randomized to same group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Right Unilateral (RUL) ECT | Bilateral (BL) ECT | Control Group
Number analyzed (Participants) | 2 | 0 | 0
units on a scale | 11.5 (3.5) |  |

2. Secondary Outcome: Depression on the Hamilton Depression Scale
Description: Repetitive evaluation by the Hamilton depression scale - To measure efficacy of ECT
Time Frame: 30 days
Population: Data not collected
Arm/Group | Right Unilateral (RUL) ECT | Bilateral (BL) ECT | Control Group
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Cognitive Side Effects on Montreal Cognitive Assessment (MoCA)
Description: Repetitive evaluation by the Montreal Cognitive Assessment (MoCA)- To evaluate possible cognitive side effects.
Time Frame: 30 days
Population: Data not collected
Arm/Group | Right Unilateral (RUL) ECT | Bilateral (BL) ECT | Control Group
Number analyzed (Participants) | 0 | 0 | 0

4. Primary Outcome: Catatonia on the Bush- Francis Scale (BFCRS) - Pre
Description: as for outcome 1
Time Frame: 1 day post first ECT treatment
Population: Only two participants enrolled because study ended. Both randomized to same group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Right Unilateral (RUL) ECT | Bilateral (BL) ECT | Control Group
Number analyzed (Participants) | 2 | 0 | 0
units on a scale | 5 (1) |  |

ADVERSE EVENTS:
Time Frame: AE data collected over a period of 8 days for one patient and a period of 3 days for the other patient during each patient's participation in the study.
Description: Only two participants were enrolled and they were both in the RUL arm of the study, so there were no patients at risk in either of the other arms.
Arm/Group | Right Unilateral (RUL) ECT | Bilateral (BL) ECT | Control Group
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/2 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This study was terminated in December 2018 because it was too difficult to enroll. Participants did not complete all the assessments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/98/NCT02734498/Prot_SAP_000.pdf